CLINICAL TRIAL: NCT07294651
Title: Effectiveness of Different Percutaneous Electrolysis Treatment Protocols Targeting the Upper Trapezius Muscle in Chronic Neck Pain: A Randomized Controlled Trial
Brief Title: Percutaneous Electrolysis of the Upper Trapezius in Chronic Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sivas State Hospital (Other)
Responsible Party: Principal Investigator, Serkan Polat, MD, Sivas State Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPTE-MAS-001-S
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Myofascial Pain of Upper Trapezius Muscle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Intensity Percutaneous Electrolysis of the Upper Trapezius plus Exercise (Active Comparator): Participants receive a home-based stretching exercise program targeting the upper trapezius muscle, plus three sessions of ultrasound-guided percutaneous electrolysis applied to the active myofascial trigger points of the upper trapezius muscle on days 1, 8, and 14. Percutaneous electrolysis is delivered using 0.3-mm acupuncture needles and an EPTE® percutaneous electrolysis device with a low-intensity protocol (0.5 mA for 90 seconds per session).
  Interventions:
  Low-Intensity Percutaneous Electrolysis of the Upper Trapezius
  Upper Trapezius Stretching Exercise Program
  Interventions: Device: Low-Intensity Percutaneous Electrolysis of the Upper Trapezius; Other: Upper Trapezius Stretching Exercise Program
- High-Intensity Percutaneous Electrolysis of the Upper Trapezius plus Exercise (Experimental): Participants receive the same home-based stretching exercise program targeting the upper trapezius muscle as the active comparator group, plus three sessions of ultrasound-guided percutaneous electrolysis applied to the active myofascial trigger points of the upper trapezius muscle on days 1, 8, and 14. Percutaneous electrolysis is delivered using 0.3-mm acupuncture needles and an EPTE® percutaneous electrolysis device with a high-intensity protocol (3 mA for 3 seconds, repeated 3 times per session).
  Interventions:
  High-Intensity Percutaneous Electrolysis of the Upper Trapezius
  Upper Trapezius Stretching Exercise Program
  Interventions: Device: High-Intensity Percutaneous Electrolysis of the Upper Trapezius; Other: Upper Trapezius Stretching Exercise Program

INTERVENTIONS:
Device: Low-Intensity Percutaneous Electrolysis of the Upper Trapezius — Ultrasound-guided percutaneous electrolysis applied to the active myofascial trigger points of the upper trapezius muscle using 0.3-mm acupuncture needles and an EPTE® percutaneous electrolysis device. A low-intensity protocol is used (0.5 mA for 90 seconds per session) on days 1, 8, and 14.
  Arms: Low-Intensity Percutaneous Electrolysis of the Upper Trapezius plus Exercise
Device: High-Intensity Percutaneous Electrolysis of the Upper Trapezius — Ultrasound-guided percutaneous electrolysis applied to the active myofascial trigger points of the upper trapezius muscle using 0.3-mm acupuncture needles and an EPTE® percutaneous electrolysis device. A high-intensity protocol is used (3 mA for 3 seconds, repeated 3 times per session) on days 1, 8, and 14.
  Arms: High-Intensity Percutaneous Electrolysis of the Upper Trapezius plus Exercise
Other: Upper Trapezius Stretching Exercise Program — Home-based stretching exercise program targeting the upper trapezius muscle throughout the treatment period in both groups.

SUMMARY:
In the planned study, we aim to investigate the effectiveness of percutaneous electrolysis treatment applied to myofascial trigger points in the upper trapezius muscle in patients with chronic neck pain. Two different protocols, a low-intensity (0.5 mA × 90 s) and a high-intensity (3 mA × 3 s × 3 repetitions), will be compared in the study.

Patients participating in the research will be randomized into 2 groups using a computer program. Stretching exercises targeting the upper trapezius muscle will be given to both groups as a home exercise program. In both groups, the percutaneous electrolysis treatment protocol will be performed on the active myofascial trigger points in the upper trapezius muscle on the 1st, 8th, and 14th days of treatment, using 0.3-millimeter acupuncture needles and an EPTE® percutaneous electrolysis device (Ionclinics & A. Deionic SL, Valencia, Spain). The low-intensity (0.5 milliampere × 90 s) treatment protocol will be applied to Group 1, and the high-intensity (3 milliampere × 3 s × 3 repetitions) treatment protocol will be applied to Group 2. In the study, two different protocols, low-intensity (0.5 mA × 90 s) and high-intensity (3 mA × 3 s × 3 repetitions), will be compared. In this way, it is aimed both to obtain information about optimal dosing and to contribute to the literature for a frequently involved muscle such as the upper trapezius.

ELIGIBILITY:
Inclusion Criteria:

Patients who agree to participate in the study, are between 18 and 70 years of age, have had symptoms for at least 3 months, and have chronic neck pain with active myofascial trigger points in the upper trapezius muscle will be included.

Exclusion Criteria:

Patients with malignancy, active infection, a history of widespread inflammatory rheumatic disease or fibromyalgia, trauma, skin lesions, infection or open wounds at the myofascial trigger point region, coagulopathy, warfarin use, a history of spinal or shoulder disorders, previous neck or upper extremity surgery, acute illness, muscle diseases, epilepsy, use of sedative medications, needle phobia, previous dry needling treatment for myofascial pain, a cardiac pacemaker, metal implants in the treatment area, conditions that contraindicate physiotherapy such as pregnancy, or metal allergy will not be included in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity (VAS) | Baseline (before treatment), immediately after completion of the 3rd treatment session (approximately 2 weeks), and 3 months after treatment initiation.
  Pain intensity related to plantar heel pain will be assessed using a 10-cm Visual Analog Scale (VAS). Higher scores indicate greater pain.

SECONDARY OUTCOMES:
Change in Pressure Pain Threshold (Algometry) | Baseline, post-treatment (approximately 2 weeks), and 3 months after treatment initiation.
  Pressure will be applied with an algometer at a right angle to the point on the plantar fascia where tenderness is most pronounced, and the patient will be asked to indicate the level at which discomfort is felt. The pressure value at which pain occurs will be determined as the pain threshold, and the pressure-pain threshold will be objectively assessed and recorded. Measurements will be repeated three times, and the best value will be recorded.
Change in Functional Disability (Modified Neck Disability Index) | Baseline (prior to the first treatment session), immediately after completion of treatment (after the third session, approximately 2 weeks from baseline), and 3 months after treatment initiation.
  Functional disability related to neck pain will be assessed using the Modified Neck Disability Index (MNDI), a 10-item questionnaire evaluating pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. Each item is scored from 0 to 5, yielding a total score between 0 and 50; higher scores indicate greater disability. The validated Turkish version of the scale will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Sivas Devlet Hastanesi, Sivas, Turkey (Türkiye)